CLINICAL TRIAL: NCT06178861
Title: Effect of Bra Use During Radiotherapy for Breast Cancer Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hwa Kyung Byun, professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9-2023-0052
Record Dates: First submitted 2023-12-04; First posted 2023-12-21 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Radiation Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Test group: Group wearing a radiotherapy bra / Control group: Group not wearing a radiotherapy bra -Allocation: Random -Blinding: None -Time: Prospective
Masking Description: Test group: Group wearing a radiotherapy bra / Control group: Group not wearing a radiotherapy bra -Allocation: Random -Blinding: None -Time: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group wearing a bra (Experimental): Patients wear a bra while receiving radiotherapy.
  Interventions: Device: Group wearing a radiotherapy bra
- Group not wearing a bra (No Intervention): Patients do not wear a bra while receiving radiotherapy.

INTERVENTIONS:
Device: Group wearing a radiotherapy bra — Group wearing a radiotherapy bra
  Arms: Group wearing a bra

SUMMARY:
This prospective randomized study investigated the reproducibility of breast shape, radiation dose irradiated to the lungs, heart, dose distribution, patient satisfaction, and treatment toxicity when wearing and not wearing a bra during radiotherapy for patients with breast cancer.

DETAILED DESCRIPTION:
Post-surgery radiotherapy to the breast is standard treatment after breast-conserving surgery in patients with breast cancer. In order to apply the latest radiation therapy technologies, such as intensity-modulated radiotherapy, it is important to maintain the correct posture. However, due to the nature of the breast made of soft tissue, it is difficult to maintain the same breast shape during each treatment. This is especially difficult for large, ptotic breasts. Accordingly, we developed a bra for breast cancer patients in order to perform accurate radiotherapy. It was designed to fix the breast using bands in various directions so that its shape and position can be fixed during radiation treatment.

This is a prospective, randomized controlled study to evaluate the effects of using a bra for breast cancer patients on the reproducibility of breast shape, radiation dose irradiated to the lungs, heart, dose distribution, patient satisfaction, and treatment toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed invasive breast cancer or ductal carcinoma in situ
2. Patients eligible for whole breast irradiation after partial mastectomy
3. Adults over 20 years old
4. Patients with good overall performance (ECOG PS 0-1)

Exclusion Criteria:

1. Recurrent breast cancer patients
2. Patients who have previously received radiation therapy to the ipsilateral breast
3. Patients who underwent breast reconstruction
4. Bilateral breast cancer
5. Patients with skin diseases such as contact dermatitis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — breast cancer
Enrollment: 38 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
The reproducibility of breast shape through cross-correlation values, both with and without the use of a bra | During the radiotherapy, an average of 1 month
  Evaluating the reproducibility of breast shape through cross-correlation values in cone-beam CT and planning CT matching. This study involves comparing groups of patients wearing and not wearing a bra

SECONDARY OUTCOMES:
Radiation dosimetric evaluation | at the time of completion of radiotherapy
  radiation dose to lungs, heart and breast
Patient satisfaction assessment | at the time of completion of radiotherapy
  1. Survey on anxiety before and after radiation treatment (using STAI, APAIS, and LASA scales)
  2. Survey on satisfaction with radiotherapy bra after radiation therapy
Assessment of treatment toxicity | at 6 months and 12 months after the radiotherapy
  1. Acute toxicity grade 2 or higher according to CTCAE version 5.0
  2. Late toxicity grade 2 or higher according to CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Hwakyung BYUN, professor, Principal Investigator — Severance Hospital
Locations (1):
- Yongin Severance Hospital, Yongin-si, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Byun HK, Kim H, Son J, Cho Y, Kwon YJ, Kim DW, Lee H, Kim YB. Impact of bra application in breast cancer radiotherapy: A pilot prospective randomized trial. Radiother Oncol. 2025 May;206:110785. doi: 10.1016/j.radonc.2025.110785. Epub 2025 Feb 12. PMID 39952437